CLINICAL TRIAL: NCT00572247
Title: The Intervention Involves Education on Nutrition and Physical Activity. Outcomes Evaluate Changes in BMI.
Brief Title: The Psychiatric Rehabilitation Approach to Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1R34MH077282-01A1 (NIH); 10575
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Schizophrenic Disorders
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Behavioral
  Interventions: Behavioral: Psychiatric Rehabilitation Approach to Weight Loss
- 2 (No Intervention)

INTERVENTIONS:
Behavioral: Psychiatric Rehabilitation Approach to Weight Loss — The use of psychiatric rehabilitation as a way to lose weight
  Arms: 1

SUMMARY:
The primary aim of the project is to examine the efficacy of the Psychiatric Rehabilitation Weight Loss program in reduction of weight and body mass index (BMI.

DETAILED DESCRIPTION:
The study involves 144 individuals who will be randomly assigned to the intervention group or treatment as usual group(control group). All Participants will undergo baseline assessment, assessment at week 12, week 24 and in year from baseline.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of serious mental illness,
* Age 18 - 65
* BMI > 25
* Medication stable (there have been no changes in antipsychotic medications or mood stabilizers for the last 3 months).

Exclusion Criteria:

* Current or history of eating disorder
* Pregnant or breast feeding
* Uncontrolled HTN
* Severe coronary artery disease
* Severe valvular disease
* Uncontrolled diabetes
* Sustained arrhythmia
* Insulin using severe physical limitations
* Severe Lung Disorders
* Diagnosis of MR or dementia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2007-01; Primary Completion 2010-01 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The reduction of weight and Body Mass Index (BMI) | Week 12, Week 24, 1 Year from Baseline Visit

SECONDARY OUTCOMES:
Measure of waist circumference, health promotion practices, dietary intake assessment of physical activity | Baseline, 12 Weeks, 24 weeks, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Edna Hamera, PhD, RN, CS, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States